CLINICAL TRIAL: NCT02748525
Title: Evaluation of Gallbladder Contractility Using Both CCK and Milk Consecutively
Acronym: Milk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Isis W Gayed, Associate Professor of Radiology - Clinical, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-16-0015
Record Dates: First submitted 2016-04-04; First posted 2016-04-22 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — Milk; Cholecystokinin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CCK then Milk (Experimental): CCK administered and HIDA scan performed. Results analyzed, if ejection fraction is low, patient is given milk to drink, and HIDA scan performed again. Results are analyzed to determine if ejection fraction is still low.
  Interventions: Other: Milk; Biological: CCK

INTERVENTIONS:
Other: Milk — Milk, in the form of 8 oz. half and half, administered after CCK scan, and patient is rescanned and ejection fraction measured to determine if ejection fraction is low.
Biological: CCK — CCK is standard of care, used in HIDA scans for gallbladder function evaluation. It is given intravenously to cause the gallbladder to contract. The usual dose of CCK is 0.02mg/kg slowly over 3 minutes as per standard.
  Other Names: Cholecystokinin

SUMMARY:
This study aims to combine the use of IV CCK administration followed by oral milk during a HIDA scan to further stimulate the gallbladder contractility and decrease the number of false abnormal HIDA scans and unnecessary cholecystectomies in some patients.

DETAILED DESCRIPTION:
Hepatobiliary imaging (HIDA) has an important role in the evaluation of the function and dynamics of the hepatobiliary system and the flow of bile to the gastrointestinal system. Contractility of the gallbladder is one of the functions that are uniquely evaluated using a HIDA scan. Poor contractility of the gallbladder can be the source of pain in many patients. Anatomic imaging studies like ultrasound, CT and/or MRI are usually normal in these patients.

Contractility of the gallbladder is evaluated during a HIDA scan by intravenous injection of cholecystokinin (CCK) a physiologic peptide enzyme produced in the duodenum in response to the presence of fatty meal which causes the gallbladder to contract and the sphincter of Oddi to relax, thus allowing the flow of bile from the gallbladder to the duodenum. CCK is usually administered during a HIDA scan intravenously after filling of the gallbladder with radioactive tracer to simulate the action of the endogenous CCK in contracting the gallbladder and relaxation of the sphincter of Oddi. Gallbladder ejection fraction (GBEF) in response to CCK injection is calculated using special computer software program. A normal gallbladder ejection fraction is equal to or greater than 35%. Alternative to CCK injection, the patient may be administered milk as a fatty drink that should stimulate a normal gallbladder to contract when it reaches the duodenum approximately 15-20 minutes after oral administration. Thus, gallbladder contractility may be evaluated during a HIDA scan either by injecting CCK intravenously or oral administration of milk. Poor contractility of the gallbladder may result in abdominal pain usually triggered by meals. However, in many patients with abdominal pain and a decreased gallbladder contractility as evaluated by IV CCK or milk may continue to suffer from pain even after surgical removal of the gallbladder . This suggests that abnormally decreased GBEF after CCK or milk stimulation may represent false abnormal finding resulting in unnecessary cholecystectomies in some of the patients. There are no reports in the literature that have used both intravenous CCK stimulation and oral milk administration together in the same patient.

This study aims to combine the use of IV CCK administration followed by oral milk during a HIDA scan to further stimulate the gallbladder contractility and decrease the number of false abnormal HIDA scans and unnecessary cholecystectomies in some patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to a HIDA scan for evaluation of gallbladder function.
* No evidence of gallbladder stones on any prior anatomic imaging studies.
* Patients who are able to lie flat on the imaging table for an additional 30 min. of imaging after the standard of care 1.5 hour HIDA scan.

Exclusion Criteria:

* Patients who are under 18 years of age.
* Patients with evidence of gallbladder stones on other imaging modalities.
* Patient allergic to milk or dairy products.
* HIDA scan ordered to evaluate for acute cholecystitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isis W Gayed, MD, Principal Investigator — University of Texas Healtlh Science Center at Houston
Locations (1):
- University of Texas Health Science Center Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards MA, Mullenbach B, Chamberlain SM. Pain provocation and low gallbladder ejection fraction with CCK cholescintigraphy are not predictive of chronic acalculous gallbladder disease symptom relief after cholecystectomy. Dig Dis Sci. 2014 Nov;59(11):2773-8. doi: 10.1007/s10620-014-3213-4. Epub 2014 May 23. PMID 24852884
- [Background] DiBaise JK, Oleynikov D. Does gallbladder ejection fraction predict outcome after cholecystectomy for suspected chronic acalculous gallbladder dysfunction? A systematic review. Am J Gastroenterol. 2003 Dec;98(12):2605-11. doi: 10.1111/j.1572-0241.2003.08772.x. PMID 14687804
- [Background] Hadigan C, Fishman SJ, Connolly LP, Treves ST, Nurko S. Stimulation with fatty meal (Lipomul) to assess gallbladder emptying in children with chronic acalculous cholecystitis. J Pediatr Gastroenterol Nutr. 2003 Aug;37(2):178-82. doi: 10.1097/00005176-200308000-00017. PMID 12883305
- [Background] Al-Muqbel KM, Bani Hani MN, Elheis MA, Al-Omari MH. Reproducibility of gallbladder ejection fraction measured by Fatty meal cholescintigraphy. Nucl Med Mol Imaging. 2010 Dec;44(4):246-51. doi: 10.1007/s13139-010-0046-8. Epub 2010 Oct 13. PMID 24899960
- [Background] Al-Muqbel KM. Gallbladder ejection fraction measured by fatty meal cholescintigraphy: is it affected by extended gallbladder emptying data acquisition time? Ann Nucl Med. 2010 Jan;24(1):29-34. doi: 10.1007/s12149-009-0324-7. Epub 2009 Nov 25. PMID 19937405
- [Background] Delgado-Aros S, Cremonini F, Bredenoord AJ, Camilleri M. Systematic review and meta-analysis: does gall-bladder ejection fraction on cholecystokinin cholescintigraphy predict outcome after cholecystectomy in suspected functional biliary pain? Aliment Pharmacol Ther. 2003 Jul 15;18(2):167-74. doi: 10.1046/j.1365-2036.2003.01654.x. PMID 12869076

RESULTS

PARTICIPANT FLOW:
Groups:
- CCK Then Milk: cholecystokinin (CCK) administered and Hepatobiliary imaging (HIDA) scan performed. Results analyzed, if ejection fraction is low, patient is given milk to drink, and HIDA scan performed again. Results are analyzed to determine if ejection fraction is still low.
  CCK: CCK is standard of care, used in HIDA scans for gallbladder function evaluation. It is given intravenously to cause the gallbladder to contract. The usual dose of CCK is 0.02mg/kg slowly over 3 minutes as per standard.
  Milk: Milk, in the form of 8 oz. half and half, administered after CCK scan, and patient is rescanned and ejection fraction measured to determine if ejection fraction is low.
Period: Overall Study
Arm/Group | CCK Then Milk
Started | 50
Completed Study Intervention | 50
Completed | 39 (Completed 6 months follow up)
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | CCK Then Milk
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  Black | 13
  White | 19
  Other | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Gallbladder Ejection Fraction
Description: Patient will receive CCK, be scanned, and the ejection fraction will be measured.
Time Frame: 30 minutes after CCK administration
Measure: Mean (Full Range); unit: percentage of ejection of tracer
Arm/Group | CCK Then Milk
Number analyzed (Participants) | 50
percentage of ejection of tracer | 15 [0 to 33]

2. Primary Outcome: Gallbladder Ejection Fraction
Description: Patient will receive CCK, be scanned, and the ejection fraction will be measured. Then milk will be administered, repeat scan and ejection fraction will be measured.
Time Frame: 45 minutes after milk administration
Measure: Mean (Full Range); unit: percentage of ejection of tracer
Arm/Group | CCK Then Milk
Number analyzed (Participants) | 50
percentage of ejection of tracer | 30 [2 to 88]

3. Secondary Outcome: Number of Participants Who Reported Abdominal Pain at 6 Months
Description: Significant pain scale at follow up was defined as 5 or greater on a scale of 0-10, with 10 being the most severe pain.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CCK Then Milk
Number analyzed (Participants) | 39
Participants | 6

4. Secondary Outcome: Number of Participants Who Received Cholecystectomy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CCK Then Milk
Number analyzed (Participants) | 39
Participants | 18

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CCK Then Milk
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 2/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CCK Then Milk (N=50)
Abdominal Pain (Hepatobiliary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT02748525/Prot_SAP_000.pdf